CLINICAL TRIAL: NCT06357039
Title: Validation Study of an Artificial Intelligence-based Sleep Stage Classification for a Home Sleep Tracking Device
Brief Title: Validation Study of Sleep Tracking Devices
Status: Completed | Type: Observational
Sponsor: PNAPS Health Informatics and Space Technologies Inc. (Other)
Collaborators: Analog Devices (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09.2023.422; 2220124 (Other Grant/Funding Number: Scientific and Technological Research Council of Türkiye (TÜBİTAK)); 1065371 (Other Grant/Funding Number: Small and Medium Enterprises Development Organization (KOSGEB))
Record Dates: First submitted 2024-02-22; First posted 2024-04-10 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Sleep; Sleep Disorder
Keywords: Sleep; Polysomnography; EEG; PPG; Wearable Device
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Participants aged 18-65 who identify as female for biological
  Interventions: Device: Sleep tracking device
- Male: Participants aged 18-65 who identify as male for biological
  Interventions: Device: Sleep tracking device

INTERVENTIONS:
Device: Sleep tracking device — In addition to polysomnography, a device containing EEG+PPG sensors for sleep classification was placed on the forehead, and another device containing PPG and accelerometer sensors was placed on the wrist. The wrist to which the device is attached is randomly assigned.

SUMMARY:
In this study, a two-part recursive convolutional neural networks model was developed, extracting features for each epoch window independently from before and after sleep onset (epoch encoder), and then trained in the context of long-term relationships in the sleep process (sequence encoder), using an approach similar to human expert classification based on information from single-channel forehead EEG and PPG (IR, Green, Red). The classification is based on guidelines from the American Academy of Sleep Medicine and calculated six parameters: total sleep duration (TST), wake (W), N1, N2, N3, and REM.

The validation study of the developed model and the device was conducted at the Sleep Disorders Centre of the Istanbul Medical Faculty using concurrent polysomnographic data from 305 male and female patients aged 18 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants suffering from sleep disorders
* Participants sent to PSG test by neurologists, pulmonologists, psychiatrists, and otolaryngologists

Exclusion Criteria:

* Anyone who has been diagnosed as having a contagious skin disease
* Participants who do not have consent to have an additional device in their forehead area
* Incomplete of sleep measurement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals aged between 18 and 65 who have voluntarily agreed to undergo sleep measurements specifically individuals suffering from sleep disorders such as sleep apnea. Participants in the study have been referred for polysomnography (PSG) testing by neurologists, pulmonologists, psychiatrists, and otolaryngologists.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Sleep Stages Classification Accuracy | 4-5 months
  The collected EEG data were classified according to Cohen's kappa (>85), which is considered successful in the literature. Initially the open source codes YASA, tinysleepnet and attentionsleep have been implemented. These codes yielded kappa 0.64, accuracy 0.80, kappa 0.69, accuracy 0.79 and kappa 0.65, accuracy 0.78 respectively. The values obtained do not correspond to those reported in the classification articles. Subsequently, 29 participants from our own dataset were tested in these classifications as a preliminary test, with poor results. On an individual basis, the highest cappa score was 0.51. Development of our own classification system is in progress.
Interoception analysis from PPG data collected from facial skin | 4-5 months
  According to our preliminary analyses, we found that the intermediary rhythm (0.12-0.18 Hz) associated with interoception is also present in sleep patients. In one participant, for example, a value of 0.19 was obtained as a ratio of total sleep time. In addition, an intermediary rhythm is observed in all stages of sleep, including wakefulness, light sleep, deep sleep and REM.

CONTACTS AND LOCATIONS:
Overall Officials: Asuman Çevik, Master's, Study Chair — PNAPS Health Informatics & Space Technologies Inc.; Hasan Birol Çotuk, PhD, Study Director — Marmara University
Locations (1):
- Pnaps Health Informatics and Space Technologies Inc, Istanbul, Başıbüyük, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The PSG data will be shared, but the main structure is not yet planned.

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT06357039/Prot_000.pdf
  • Informed Consent Form (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT06357039/ICF_001.pdf